CLINICAL TRIAL: NCT01302496
Title: A Two-stage Phase II Study of Autologous TriMix-DC Therapeutic Vaccine in Combination With Ipilimumab in Patients With Previously Treated Unresectable Stage III or IV Melanoma
Brief Title: Autologous TriMix-DC Therapeutic Vaccine in Combination With Ipilimumab in Patients With Previously Treated Unresectable Stage III or IV Melanoma
Acronym: TriMix-Ipi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bart Neyns (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor-Investigator, Bart Neyns, MD PhD, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UZB-VUB-10-001; 2010-023058-35 (EudraCT Number)
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Malignant Melanoma Stage III; Malignant Melanoma Stage IV
Keywords: Previously Treated; Unresectable; Stage III or IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TriMix-DC and Ipilimumab (Experimental)
  Interventions: Biological: TriMix-DC and ipilimumab

INTERVENTIONS:
Biological: TriMix-DC and ipilimumab — Patients will receive 5 administrations of autologous TriMix-DC, administrations 2, 3, 4 and 5 will be preceded by ipilimumab (a CTLA-4 blocking monoclonal antibody, at a dose of 10 mg/kg). Patients who are free from progression according to the irRC will be offered ipilimumab maintenance administrations of ipilimumab (10mg/kg q12wks).

SUMMARY:
The CTLA-4 blocking monoclonal antibody ipilimumab (MDX-010, BMS-734016), has demonstrated anti-tumor activity in a subgroup of patients with Stage III (unresectable) or Stage IV melanoma (measurable per modified WHO criteria), who have received prior treatment with any regimen (non-experimental or experimental), except a CD-137 agonist or a CTLA4 inhibitor or agonist and relapsed, failed to respond (CR or PR) or did not tolerate that regimen (Wolchok, Neyns et al. 2009; O'Day, Maio et al. 2010). Ipilimumab exerts its therapeutic effect presumably by activating T-lymphocytes that infiltrate the tumor mass to destroy the malignant cells by mechanisms of cytotoxic cellular interaction. Autologous TriMix-DC vaccine can induce a T-cell repertoire that recognizes in a HLA-restricted way the melanoma associated antigens MAGE-A3, MAGE-C2, tyrosinase and gp100. Administration of ipilimumab together with TriMix-DC vaccine therapy may be a more effective treatment for patients with advanced melanoma as compared to either modality alone.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent;
2. Accessible for treatment and follow-up;
3. Histologically confirmed malignant melanoma; primary melanoma of the skin, or unknown primary site (patients with primary mucosa or uveal melanoma are not eligible).
4. Measurable melanoma, as per irRC criteria;
5. AJCC Stage III (unresectable) or Stage IV melanoma;
6. Patient must have demonstrated one of the following in response to treatment with at least one prior regimen (non-experimental or experimental) with the exception of a CD137 agonist or PD-1 or CTLA-4 inhibitor or agonist:

   * relapse following an objective response of PR or CR; or
   * failed to demonstrate an objective response of PR or CR based on an assessment period of at least 12 weeks from prior regimen start; or
   * inability to tolerate treatment due to toxicity;
7. Have a complete set of baseline (i.e., Screening) digital images of lesions and radiographic images, including, but not limited to: brain, bone, chest, abdomen and pelvis.
8. Required values for initial laboratory tests:

   WBC > 2500/mm³ ANC > 1500/ mm³ Platelets > 75 x 103/uL Hemoglobin > 9 g/dL (may be transfused) Creatinine < 2.0 x ULN AST/ALT < 2.5 x ULN for patients without liver metastasis, < 5 times for liver metastases Bilirubin < 2.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
9. No active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
10. ECOG performance status of 0 or 1;
11. Life expectancy of > 16 weeks;
12. Men and women, >= 18 years of age. The following paragraphs are mandatory when the protocol includes Women of Childbearing Potential.
13. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized. In general, the decision for appropriate methods to prevent pregnancy should be determined by discussions between the investigator and the study subject. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:

    * Amenorrhea > 12 consecutive months without another cause, or
    * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL.

    Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.

    WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.

    Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.
14. Adequate venous access allowing for a leukapheresis procedure.

Exclusion Criteria:

1. Evidence of brain metastases on brain imaging (i.e., MRI or contrast CT);
2. Primary ocular or mucosal melanoma;
3. Any other malignancy form which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
4. Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
5. Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
6. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
7. A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA 4 inhibitor or agonist, or PD-1 antagonist;.
8. Concomitant therapy with any of the following: IL 2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses);
9. Concomitant therapy with and need of uninterrupted therapeutic anticoagulation (e.g. because of a recent thrombo-embolic event or cardiac valve prothesis).
10. Previous treatment with other investigational products, including cancer immunotherapy, within 30 days preceding study recruitment;
11. Previous treatment in another ipilimumab clinical trial or prior treatment with a CD137 agonist, CTLA-4 inhibitor or agonist;
12. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness.
13. Women of childbearing potential (WOCBP), defined above in Section 4.1, who:

    * are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug, or
    * have a positive pregnancy test at baseline, or
    * are pregnant or breastfeeding. Sexually active WOCBP must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Before study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy. All WOCBP MUST have a negative pregnancy test before first receiving ipilimumab. If the pregnancy test is positive, the patient must not receive ipilimumab and must not be enrolled in the study.
14. Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 8 weeks after ipilimumab is stopped.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
disease control rate according to the immune-related response criteria | Response evaluation by PET/CT every 12 weeks following initiation of study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brabant, Belgium

REFERENCES:
- [Derived] De Keersmaecker B, Claerhout S, Carrasco J, Bar I, Corthals J, Wilgenhof S, Neyns B, Thielemans K. TriMix and tumor antigen mRNA electroporated dendritic cell vaccination plus ipilimumab: link between T-cell activation and clinical responses in advanced melanoma. J Immunother Cancer. 2020 Feb;8(1):e000329. doi: 10.1136/jitc-2019-000329. PMID 32114500